CLINICAL TRIAL: NCT03994978
Title: Preoperative vs. Postoperative Bowel Function and Quality of Life in Patients Undergoing Elective Sigmoidectomy vs. Conservative Management for Recurrent Uncomplicated Diverticulitis (FRESCO-Trial)
Brief Title: Bowel Function/QoL After Elective Sigmoidectomy vs. Conservative Management for Recurrent Uncomplicated Diverticulitis
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: FRESCO Trial
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Diverticulitis of Sigmoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical group: Patients with uncomplicated recurrent diverticulitis undergoing elective sigmoid resection
  Interventions: Procedure: elective sigmoidectomy
- Conservative group: Patients with uncomplicated recurrent diverticulitis with conservative treatment

INTERVENTIONS:
Procedure: elective sigmoidectomy — elective sigmoidectomy
  Groups: Surgical group

SUMMARY:
The decision to perform a surgical intervention or not after recovery from repeated uncomplicated episodes of acute diverticulitis remains controversial and the literature shows different conflicting approaches based on low-quality evidence.The goal of this trial is to achieve a better understanding of the impact of surgery on bowel function and QoL in patients with recurrent uncomplicated sigmoid diverticulitis in order to develop treatment guidelines.

DETAILED DESCRIPTION:
The prevalence of diverticular disease of sigmoid in the Western has increased over the past century and our know-how of this disease and its management continues to evolve. International experts have tried to standardize the surgical approach to patients with recurrent episodes of sigmoid diverticulitis but, to date, no guidelines are universally recognized.The American Society of Colon and Rectal Surgeons (ASCRS) and the World Society of Emergency Surgery (WSES) recommend an individualized approach after recovery from uncomplicated acute diverticulitis to plan an elective sigmoid resection. The impact of ongoing disorders on quality of life (QoL) and not the number of previous episodes of diverticulitis should be the most determining factor. The German guideline by the Deutsche Gesellschaft für Allgemein- und Viszeralchirurgie (DGAV) recommend an elective sigmoid resection after a careful risk/benefit assessment depending on the clinical presentation in the disease-free interval in patients with chronic relapsing diverticulitis.The Danish Surgical Society (DSS) is more restrained and mentions the unnecessary risk in terms of morbidity and mortality to the individual as well as costs to society in prophylactic resection of the sigmoid. Therefore, they recommend that elective surgery should be probably limited to symptomatic cases not amenable to conservative measures. Moreover, recent studies have demonstrated that the number of attacks of diverticulitis is not necessarily a prevailing factor in defining the suitability of surgery and the operation itself carries significant morbidity and mortality. The German guidelines describe also a persistence of the symptoms in patients who underwent sigmoid resection in 22-25%. An uncomplicated diverticulitis is generally considered a mild and self-limiting disease, performing a potentially harmful procedure in these patients does not seem justified. However, elective resection may be an appropriate solution for a more selective group of patients who suffer greatly from their disease. Many studies have consistently shown that 40-80% remain symptomatic after conservative treatment, leading to impaired health-related Quality of life (HRQoL) and increased costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent uncomplicated diverticulitis and surgical indication for sigmoid resection
* Patients with recurrent uncomplicated diverticulitis and non-surgical indication for conservative management
* Confirmation of at least one episode of acute uncomplicated diverticulitis in computed tomography

Exclusion Criteria:

* Patients aged under 18.
* Patients unable to understand an informed consent.
* Patients with chronic pain disorder.
* Patients with sigmoid fistulas
* Emergency operations.
* Pregnant women or lactation.
* Patients with other severe gastrointestinal diseases, such as inflammatory bowel diseases (IBD), carcinoma or immunologic disorders.
* Patients unable to perform surgery or high-risk patients according to the American Society of Anesthesiology (ASA 4 grade or higher)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent episodes of diverticulitis with indication of further treatment.The physician decides which therapy (conservative or surgical) will be carried out.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Change in grade of fecal incontinence incontinence score | change from baseline to 12 months after intervention
  Fecal incontinence measured by total "Vaizey-Wexner incontinence score" ranging from 0 to 24; lower values represent better outcome
Change in grade of constipation | change from baseline to 12 months after intervention
  Constipation measured by total "Cleveland constipation score" ranging from 0 to 30; lower values represent better outcome

SECONDARY OUTCOMES:
Change in gastrointestinal quality of Life: gastrointestinal quality of life score" (GIQLI score) | change from baseline to 12 months after intervention
  Gastrointestinal quality of life measured by total "gastrointestinal quality of life score" (GIQLI score) ranging from 0-144; higher values represent better outcome
Change in erectile function | change from baseline to 12 months after intervention
  Erectile function measured by total "international index of erectile function" (IIEF-5-score) ranging from 5 to 25; higher values represent better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Wölnerhanssen, MD, Study Chair — St. Clara Research Ltd.; Daniel Steinemann, MD, Principal Investigator — Clarunis
Locations (1):
- St. Claraspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No